CLINICAL TRIAL: NCT05466448
Title: An Open Label Phase 2 Study to Compare the Pharmacokinetics, Efficacy and Safety of RZL-012 in Chinese Subjects Seeking Submental Fat Reduction vs. Non-Chinese Subjects Seeking Submental Fat Reduction
Brief Title: An Open Label Study That Will Test Safety and Efficacy of RZL-012 Injection Into the Submental Fat in Chinese vs. Non-Chinese Subjects.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Raziel Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RZL-012-SMFC-P2US-001
Record Dates: First submitted 2022-06-16; First posted 2022-07-20 (Actual); Results first posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-11

CONDITIONS: Submental Fat
MeSH Terms: interventions — RZL-012

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RZL-012 50mg/ml (Experimental): small synthetic molecule for submental fat reduction
  Interventions: Drug: RZL-012

INTERVENTIONS:
Drug: RZL-012 — concentration of injected formulation 50 mg/mL RZL-012 of 7.5 mg/0.15 mL/injection point that results in a maximum total dose/volume of 240±30 mg/4.8±0.6 mL RZL-012

SUMMARY:
This is a Phase 2, open label study that will consist of a screening period, baseline period in which subjects will receive a single treatment session and a follow-up period. The single treatment session will consist of multiple injections of RZL-012 into the submental area under the chin. Blood samples will be collected from all subjects for PK analyses in the first 30 hours after dosing. Subjects will thereafter be monitored for safety and efficacy for at least 84 days.

DETAILED DESCRIPTION:
• RZL-012 (concentration of injected solution 50 mg/mL RZL-012) of 7.5 mg/0.15 mL/injection point that results in a total dose/volume of 240±30mg mg/4.8±0.6 mL RZL-012

Subjects treated with RZL-012 will undergo a single treatment session with 32±4 injections. The maximal number of injections will be 36 with maximal dose of 270 mg RZL-012 .

ELIGIBILITY:
Inclusion Criteria:

* Is a male or female subject between the ages of 18 and 65 years, inclusive.
* Has body mass index (BMI) between >22 kg/m2 and <40 kg/m2.
* If enrolled for Chinese arm, subjects have to be ethnically pure, i.e., Chinese passport holders with all four grandparents being Chinese.
* Has a SMF bulge that is contiguous and fits to 32±4 injections sites according to a grid with 1 centimeter (cm) distance between injection points.
* Has grade 3 to 4 of SMF as rated by both the C-CAT and S-CAT.
* Has a visible or large pocket of submental fat- according to physician global assessment.
* Has stable weight, with no fluctuation of >5 kg in the past 12 months.
* If female, is not pregnant or breastfeeding based on the following:

  1. agree to the use of highly effective contraceptive methods for at least 2 weeks before baseline until 4 weeks after the last day of study drug and a negative serum pregnancy test (ß-hCG) at screening and negative urine pregnancy test at baseline; or
  2. is of nonchildbearing potential defined as clinically infertile as the result of surgical sterilization (hysterectomy, bilateral tubal ligation, and/or bilateral oophorectomy); or
  3. is confirmed postmenopausal status (defined as either having amenorrhea for ≥ 12 consecutive months without another cause and documented serum follicle-stimulating hormone (FSH) level > 40 mIU/mL or another documented medical condition (e.g., was born without a uterus))
* If male (with or without vasectomy), agree to the use of highly effective contraceptive methods as listed above in criteria 7 as well as to use a barrier method, e.g. condom , from study check-in until 7 days after the last day of study drug.
* Is willing to avoid strenuous exercise for seven (7) days post treatment.
* Is able to adhere to the visit schedule and protocol requirements and be available to complete the study.

  12. Is willing and able to sign an Institutional Review Board (IRB) approved informed consent form (ICF) indicating that they are aware of the investigational nature of the study.

Exclusion Criteria:

* Is unable to tolerate subcutaneous injections.
* Has dysfunctional gallbladder activity (e.g., underwent cholecystectomy or cholecystitis).
* Has any uncontrolled systemic disease that is not stabilized (i.e., cardiovascular disease, mental illness).
* Has skin laxity (i.e., elastosis, skin crepiness, skin redundancy, skin draping, vertical and/or horizontal skin bands and folds, blunting of cervical mental angle, loss of opposition of skin to underlying neck structures due to skin laxity) that could obscure the evaluation and treatment of SMF.
* Has any scars, unshaven hair, tattoos, facial hair or jewelry on or near the proposed treatment area.
* Has presence of structures or confounding factors that may interfere with assessing SMF such as but not limited to enlarged submandibular salivary and/or parotid glands, micrognanthia, chin implant, soft tissue volume augmentation of chin and/or jawline, pronounced platysmal bands and deep necklace lines or presence of facial jowls that could obscure the evaluation of SMF.
* Has a fat bulge under the chin that is too large to be adequately treated by 32±4 contiguous injections on a 1cm grid .
* Has a fat bulge under the chin that is of an insufficient volume to allow 32±4 injections within a contiguous 1 cm grid.
* Has significant history or current evidence of a medical, psychological or other disorder that, in the Investigator's opinion, would preclude enrollment in the study.
* Has an active bacterial, fungal, or viral infection in the proposed treatment area.
* Has a pre-existing skin condition in the submental region that, at the Investigator's discretion, may confound evaluation or analysis.
* Has previously had treatments or surgery in the submentum, such as but not limited to, focused ultrasound, radiofrequency, cryolipolysis, liposuction, sodium deoxycholate, or neck lift.
* Has pre-existing neurological or gastrointestinal condition leading to dysphagia, dysphonia, or facial nerve palsy.
* Has Dercum's Disease.
* Has allergic reactions to injectables.
* Has any pre-existing medical condition other than increased SMF that, at the Investigator's discretion, may result in increased submental fullness, such as but not limited to, thyroid enlargement, goiter, cervical lymphadenopathy, etc.
* Has a planned fat reduction procedure of any variety to the submental region for the duration of the study.
* Has medication or a history of coagulopathy.
* Has a history or family history of venous thrombotic disease.
* Has been treated chronically at least three (3) months prior to study entry with systemic steroids or immunosuppressive drugs.
* Has been treated chronically at least one (1) week prior to study entry with non-steroidal anti-inflammatory drugs (NSAIDs)
* Has used anticoagulation therapies that may increase bleeding or bruising (i.e., aspirin, ibuprofen, warfarin, vitamins, and herbal preparations) for seven (7) days prior to treatment.
* Has had treatment with botulinum toxin injections in the neck or chin area within 9 months prior to screening.
* Current participation or participation within three (3) months prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Luxurgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Chinese; Non-Chinese: RZL-012 50mg/ml small synthetic molecule for submental fat reduction
  RZL-012: concentration of injected formulation 50 mg/mL RZL-012 of 7.5 mg/0.15 mL/injection point that results in a maximum total dose/volume of 240±30 mg/4.8±0.6 mL RZL-012
Period: Overall Study
Arm/Group | Chinese | Non-Chinese
Started | 6 | 9
Completed | 5 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chinese | Non-Chinese | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (14.7) | 43.8 (11.9) | 40.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 0 | 7 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Measure - Drug Concentration in the Blood (ng/mL)
Description: Measurement of maximum drug concentration (Cmax) (ng/mL)
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: concentration (ng/ml)
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 6 | 9
concentration (ng/ml) | 487.7 (183.6) | 473.3 (186.8)

2. Primary Outcome: Pharmacokinetics Measure - Area Under the Plasma Concentration Versus Time Curve (AUC) (mg*h/L)
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: AUC to Last Nonzero Conc (mg*h/L)
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 6 | 9
AUC to Last Nonzero Conc (mg*h/L) | 4574.4 (987.7) | 4718.0 (1345.1)

3. Secondary Outcome: Efficacy -Change in Score According to Clinician Chin Assessment Tool (C-CAT)
Description: To determine the efficacy of RZL-012 versus placebo on submental fat (SMF) reduction measured on Day 84 versus baseline using the Clinician Chin Assessment Tool (C-CAT) by proportion of subjects with reduction in C-CAT score. The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 5 | 9
Participants | 4 | 7

4. Secondary Outcome: Efficacy - Change in Score According to Subject Chin Assessment Tool (S-CAT)
Description: To determine the efficacy of RZL-012 versus placebo on submental fat (SMF) reduction measured on Day 84 versus baseline using the Subject Chin Assessment Tool (S-CAT) by proportion of subjects who has reduction in S-CAT score. The CAT is composed of 5 points where 0 represents no fat and 4 represent very noticeable bulge and fat that extends beyond the neck
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 5 | 9
Participants | 4 | 7

5. Secondary Outcome: Efficacy - Change in Submental Fat Thickness
Description: Change from baseline in submental fat thickness (%), as measured with MRI in RZL-012 treated subjects vs. placebo treated subjects on Day 84 following injection
Time Frame: 84 days
Measure: Mean (Standard Deviation); unit: percentage of thickness reduction
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 5 | 9
percentage of thickness reduction | -34.3 (17.2) | -24.6 (23)

6. Secondary Outcome: Safety - Adverse Events Follow up
Description: To evaluate the safety of RZL-012 subcutaneous injections in the submental area in Chinese vs. non Chinese population, as assessed by spontaneous adverse event reports and post injection evaluation of treatment area. Treatment area evaluations including, but not limited to evaluation of edema, bruising, dysphasia, dysphonia, erythema, dyspigmentation, induration, numbness, pain, paresthesia, and pruritus. The number of subjects with treatment-related adverse events will be compared within each treatment group, as assessed by CTCAE v4.0
Time Frame: 84 days
Measure: Count of Participants; unit: Participants
Arm/Group | Chinese | Non-Chinese
Number analyzed (Participants) | 6 | 9
Participants | 6 | 9

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Chinese | Non-Chinese
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chinese (N=6) | Non-Chinese (N=9)
Dysphagia (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 7
Injection site haemorrhage (General disorders) | 2 | 5
Injection site hypoaesthesia (General disorders) | 0 | 4
Injection site edema (General disorders) | 6 | 9
Injection site pain (General disorders) | 6 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Skin induration (Skin and subcutaneous tissue disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT05466448/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/48/NCT05466448/SAP_001.pdf